CLINICAL TRIAL: NCT00238745
Title: Bone Mineral Density Increase and Safety of TSE-424 Compared to Placebo in Osteoporotic Postmenopausal Women
Brief Title: Study Evaluating Bazedoxifene Dose-Response in Japanese Patients With Postmenopausal Osteoporosis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 3068A1-207
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2007-12-20 (Estimated); Status verified 2007-12

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — bazedoxifene

INTERVENTIONS:
Drug: Bazedoxifene
Drug: Placebo

SUMMARY:
Dose-response in Japanese patients with postmenopausal osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* Must be postmenopausal and diagnosed as osteoporosis based on bone mineral density and/or vertebral fracture.

Exclusion Criteria:

* Diseases which possibly induce secondary osteoporosis or osteopenia and affect on bone metabolism.

Max Age: 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 375
Dates: Start 2003-08; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Bone mineral density of lumbar spine (L1-L4) at 2 years.

SECONDARY OUTCOMES:
Bone metabolic makers, bone fracture, bone mineral density of lumbar spine (L2-L4) and lip, lipid parameters, height and adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer

REFERENCES:
- [Derived] Itabashi A, Yoh K, Chines AA, Miki T, Takada M, Sato H, Gorai I, Sugimoto T, Mizunuma H, Ochi H, Constantine GD, Ohta H. Effects of bazedoxifene on bone mineral density, bone turnover, and safety in postmenopausal Japanese women with osteoporosis. J Bone Miner Res. 2011 Mar;26(3):519-29. doi: 10.1002/jbmr.252. PMID 20839291